CLINICAL TRIAL: NCT04931524
Title: An Open Label, Single-Dose Study to Assess the Mass Balance Recovery, Metabolism and Excretion of [14C] ANG 3777 in Healthy Male Subjects
Brief Title: A Study to Assess the Absorption, Metabolism and Excretion of [14C]-ANG-3777
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14C-ANG3777-HV4-102
Record Dates: First submitted 2021-05-28; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized study. Blinding is not required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- carbon-14-[14C]-ANG-3777 (Experimental): Administered IV as a single dose over 30 minutes on the morning of Day 1 following an 8 hour overnight fast and remain in the clinical unit until up to 168 hours after dosing (to Day 8). If mass balance criteria have not been met on Day 8, the clinical unit residency may be extended up to an additional 96 hours (to Day 12).
  Interventions: Drug: carbon-14-[14C]-ANG-3777

INTERVENTIONS:
Drug: carbon-14-[14C]-ANG-3777 — Arms assigned to this intervention will receive 240 mg, IV and not more than 5.2 MBq, Fasted
  Other Names: Hepatocyte growth factor mimetic

SUMMARY:
The purpose of this study is to assess the mass balance recovery and metabolic profiling and identification of 14C-ANG-3777 administered as a single IV dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 30 to 65 years inclusive at the time of signing informed consent
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 and weighing 50 to 120 kg as measured at screening
4. Must be willing and able to communicate and participate in the whole study
5. Must have regular bowel movements (ie average stool production of ≥1 and ≤3 stools per day)
6. Must provide written informed consent
7. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
2. Subjects who are, or are immediate family members of, a study site or sponsor employee
3. Evidence of current SARS-CoV-2 infection.
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
6. A confirmed positive alcohol breath test at screening or admission
7. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity (TR) in all excreta urine: CumAe and Cum%Ae | Day 1 to Day 8 (or Day 1 to Day 12)
Mass balance recovery of total radioactivity (TR) in all excreta faeces: CumAe and Cum%Ae | Day 1 to Day 8 (or Day 1 to Day 12)
Collection of plasma samples for metabolite profiling, structural identification, and quantification analysis | Day 1 to Day 8, or up to Day 12 (except for metabolite profiling up to Day 2)
Collection of urine samples for metabolite profiling, structural identification, and quantification analysis | Day 1 to Day 8, or up to Day 12 (except for metabolite profiling up to Day 2)
Collection of faeces samples for metabolite profiling, structural identification, and quantification analysis | Day 1 to Day 8, or up to Day 12 (except for metabolite profiling up to Day 2)
Determination of routes of elimination of [14C]-ANG-3777 by Ae, %Ae, CumAe and Cum%Ae by interval | Day 1 to Day 12
Determination of rates of elimination of [14C]-ANG-3777 by Ae, %Ae, CumAe and Cum%Ae by interval | Day 1 to Day 12
Measurement of the appropriate PK parameters of parent ANG-3777 in plasma including but not limited to: Tmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in plasma including but not limited to: Cmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in plasma including but not limited to: AUC(0-last) and AUC(0-inf) | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in urine including but not limited to: Tmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in urine including but not limited to: Cmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in urine including but not limited to: AUC(0-last), and AUC(0-inf) | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in faeces including but not limited to: Tmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in faeces including but not limited to: Cmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of parent ANG-3777 in faeces including but not limited to: AUC(0-last), and AUC(0-inf) | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in plasma including but not limited to: Tmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in plasma including but not limited to: Cmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in plasma including but not limited to: AUC(0-last), and AUC(0-inf) | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in urine including but not limited to: Tmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in urine including but not limited to: Cmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in urine including but not limited to: AUC(0-last), and AUC(0-inf) | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in faeces including but not limited to: Tmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in faeces including but not limited to: Cmax | Day 1 to Day 8
Measurement of the appropriate PK parameters of TR in faeces including but not limited to: AUC(0-last), and AUC(0-inf) | Day 1 to Day 8
Evaluation of whole blood:plasma concentration ratios for TR | Plasma from Day 1 to Day 8; whole blood up to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences - Nottingham, UK
Locations (1):
- Quotient Sciences, Nottingham, Nottinghamshire, United Kingdom